CLINICAL TRIAL: NCT03223103
Title: Phase I Study of Tumor Treatment Fields and a Personalized Mutation-derived Tumor Vaccine in Patients With Newly Diagnosed Glioblastoma (GCO 17-0566)
Brief Title: Safety and Immunogenicity of Personalized Genomic Vaccine and Tumor Treating Fields (TTFields) to Treat Glioblastoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Adilia Hormigo (Other)
Collaborators: NovoCure Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Adilia Hormigo, Professor, Albert Einstein College of Medicine
Organization: Albert Einstein College of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-13817; 16-089 (Other: PRMC)
Record Dates: First submitted 2017-07-18; First posted 2017-07-19 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Glioblastoma
Keywords: Brain cancer; Glioblastoma; Personalized vaccine; Polyinosinic-polycytidylic acid (Poly-ICLC); Immunotherapy; Cancer; NovoTTF-200A; Optune; GBM; immunogenicity
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Neoplasms | interventions — poly ICLC; Peptides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Mutation-derived tumor vaccine (Experimental): MTA-based Personalized Vaccine (peptides + Poly-ICLC with Tumor Treating Fields
  Interventions: Drug: Poly-ICLC; Device: Tumor Treating Fields; Biological: Peptides

INTERVENTIONS:
Drug: Poly-ICLC — Poly-ICLC 100mcg per peptide per dose
  Other Names: Hiltonol®
Device: Tumor Treating Fields — an FDA approved treatment for patients with recurrent GBM and newly diagnosed GBM
  Other Names: Optune®
Biological: Peptides — synthetic long peptides (SLP) as vaccine substrate
  Other Names: Personalized peptides

SUMMARY:
The purpose of this study is to use precision medicine in the form of a vaccine, a mutation-derived tumor antigen vaccine (MTA-based vaccine) in combination with standard care treatment of glioblastoma (GBM) and Tumor Treating Fields (TTFields).

The study is designed to determine whether this treatment combination is well tolerated and safe.

DETAILED DESCRIPTION:
This is a single-arm, single institution phase 1a / 1b study to test the safety, tolerability, and immunogenicity of MTA-based personalized vaccine in patients with newly diagnosed GBM along with the use of continual TTFields. MTA-based personalized vaccine is prepared in the laboratory with several peptides based on each patient's own tumor sequence.

The vaccine is given after the radiation and chemotherapy portion of the treatment, in the maintenance phase of temozolomide in conjunction with the TTFields.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Histological confirmation of GBM (WHO grade IV).
* Stable disease after treatment of radiation with concurrent chemotherapy. If the disease is not stable or progresses while in the study the patient is allowed to continue the study receiving the vaccine if the tumor gets controlled by other modality treatment(s)
* Must have received maximal debulking surgery and undergo radiotherapy concomitant with Temozolomide (45-70Gy)
* Life expectancy > 16 weeks
* Performance status of 0-2 as determined by Eastern Cooperative Oncology Group (ECOG) and/or Karnofsky Performance Status (KPS) 70-100
* First vaccine treatment start date at least 4 weeks out but not more than 8 weeks from the last dose of concomitant Temozolomide or radiotherapy
* Must have archival tumor tissue that is sufficient quantity and quality for sequencing
* Have adequate bone marrow function
* Requires Dexamethasone ≤ 4mg daily on a stable dose
* Acceptable hematologic, hepatic, and renal function and these tests must be performed within 14 days prior to study
* Must be deemed competent to give informed consent
* Must agree to use two effective forms of contraception beginning at least four (4) weeks prior to study entry, and continuing to do so for the duration of participation in the study

Exclusion Criteria:

* Progression of disease at time of screening
* Implanted pacemaker, programmable shunts, defibrillator, deep brain stimulator, other implanted electronic devices in the brain, or documented clinically significant arrhythmias
* Infra-tentorial tumor or multifocal disease
* History of hypersensitivity reaction to Temozolomide or a history of hypersensitivity to Decarbazine (DTIC)
* Receiving any other investigational agents. Patient is allowed to get another investigational agent and to continue receiving the vaccine only if the disease progresses while in the study and the other investigational agent is a reasonable choice to treat the patient
* Active cancer at the time of screening
* Prior history of unrelated neoplastic disease, and having received systemic therapy for the secondary malignancy within the twelve (12) month period preceding the screening evaluation.
* History of Human Immunodeficiency Virus/Acquired Immunodeficiency Syndrome (HIV/AIDS), chronic hepatitis B or hepatitis C or is otherwise reasonably suspected to meet criteria for the diagnosis of a known congenital or acquired disorder causing systemic immunosuppression
* History of, or is reasonably suspected to meet criteria for the diagnosis of a known congenital or acquired disorder causing systemic immunosuppression; or the subject is currently receiving any drug or supplement which is known to be associated with systemic immune suppression including those drugs which are prescribed for solid organ or stem cell transplant, autoimmune/inflammatory disorders, or other related medical conditions
* History of, or is reasonably suspected to meet criteria for the diagnosis of a systemic auto-immune/inflammatory disease or other autoimmune disorder with the exception of: Vitiligo, diabetes, or thyroid dysfunction
* Less than 18 years of age, or otherwise unable to give informed consent due to minor status
* Prisoner, as defined by [45 CFR 46.303(c)]
* Cognitively impaired, and unable to give informed consent
* Pregnant, as defined by a presumptive sign of pregnancy such as missed menses or a positive pregnancy test [45 CFR 46.203(b)]
* Requires or is likely to require more than a 2-week course of corticosteroids of >4mg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2029-05-12 (Estimated); Study Completion 2029-05-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLT) | long term, up to 10 years after treatment initiation
  Safety and Tolerability of the personalized treatment regimen will be assessed in tandem using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.03. NCI-CTCAE is a standard system for grading and reporting adverse events (AEs) in cancer clinical trials to document the occurrence and severity of AEs, with grades ranging from 1 (mild) to 5 (death). DLTs will be summarized and reported.
Feasibility of Personalized MTA vaccine administration | Up to 42 weeks after treatment initiation
  Feasibility of the personalized MTA vaccine will be defined as the successful administration of at least one (1) dose to subjects following tissue sample acquisition and will be expressed as the proportion or percentage subjects enrolled in the study who have successfully been administered at least one dose of the personalized MTA vaccine.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 6 months after diagnosis
  PFS will be determined by the percentage of patients whose disease remains stable, without disease progression or death, from the time diagnosis until 6 months after diagnosis.
Overall Survival (OS) | 1 year, 2 years, 5 years, and 10 years after diagnosis
  Overall Survival will be determined by from the time of diagnosis to the time of death, or up to 10 years. OS will be summarized as the percentage of patients who reach the 1-year, 2-year, 5-year, and 10-year milestones.

OTHER OUTCOMES:
Overall Response | 2 years after treatment initiation
  Overall Response will be determined as measured by Immunotherapy Response Assessment in Neuro-oncology (iRANO) criteria. Response Criteria will be summarized as either: Complete response, Partial response, Stable Disease, or Progressive Disease. The number/percentage of patients with each response type will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Adilia Hormigo, MD, PhD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided